CLINICAL TRIAL: NCT04072341
Title: Effects of Green Propolis Extract (EPP-AF) on Inflammation in Hemodialysis Patients: a Randomized Cross-over Trial.
Brief Title: Effects of Green Propolis Extract (EPP-AF) on Inflammation in Hemodialysis Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Hospital Sao Rafael (Other); Alagoas State University of Health Science , Maceió , Brazil. (Unknown)
Responsible Party: Principal Investigator, Marcelo Augusto Duarte Silveira, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Hospital São Rafael S.A
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Inflammation; Propolis; High-sensitivity C-reactive protein; Hemodialysis
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, proof-of-concept, single-center. Each patient served as their own control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis Period (Experimental): Hemodialysis patients will be under regular treatment of their comorbidities and using Propolis.
  Interventions: Drug: Propolis Period (Green Propolis 250mg/day)
- Control Period (Experimental): Hemodialysis patients will be under regular treatment of their comorbidities, but without using Propolis.
  Interventions: Other: Control Period

INTERVENTIONS:
Drug: Propolis Period (Green Propolis 250mg/day) — Randomized, cross-over, open-label. Patients will go through two 4 week periods with 1 week washout between them. During the intervention period will use 250mg of green Propolis per day. In the control period they will only follow standard treatment for their comorbidities.
  Other Names: Standard treatment for their comorbidities.
  Arms: Propolis Period
Other: Control Period — In the control period they will only follow standard treatment for their comorbidities.
  Other Names: Standard treatment for their comorbidities.
  Arms: Control Period

SUMMARY:
End-stage chronic kidney disease is associated with the condition of chronic inflammation. Patients on hemodialysis are known to be predisposed to several factors that predispose to inflammation: dialysis membranes, central venous catheters, oxidative stress, fluid overload, sodium overload, uraemic toxins. Propolis, a natural resin produced by bees from plant materials, has anti-inflammatory, immunomodulatory, and anti-oxidant properties. The aim of this study was to evaluate the impact of Brazilian green propolis extract on inflammation in hemodialysis patients.

DETAILED DESCRIPTION:
Randomized open-label cross-over trial to investigate impact of Brazilian green propolis extract on inflammation in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Male or female on hemodialysis for at least 1 month.

Exclusion Criteria:

* Pregnant Woman;
* Carriers of active neoplasms;
* Patients undergoing kidney transplantation during the study;
* Infection during the study;
* Patients who underwent parathyroidectomy during the study;
* Patient using immunosuppressive drugs;
* Allergy to propolis or any of its components;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in serum level of High-sensitivity C-reactive protein from baseline to end of study periods. | 8 weeks
  Change in high sensitivity C-reactive protein from baseline to end of study periods.

SECONDARY OUTCOMES:
Change in serum level of Interleukin-1 Beta from baseline to end of study periods. | 8 weeks
  Change in Interleukin-1 Beta from baseline to end of study periods.
Changes in serum level of alanine aminotransferase, aspartate aminotransferase, amylase and creatine kinase during the study, from baseline to end of study periods. | 8 weeks
  To evaluate the safety of propolis use in hemodialysis patients. Measurement of changes in serum level of alanine aminotransferase, aspartate aminotransferase, amylase and creatine kinase during the study.
Percentage of participants with adverse events during the study. | 8 weeks
  We will evaluate the presence or absence of symptoms related to the use of propolis through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Silveira, MD, PhD, Principal Investigator — Hospital São Rafael S.A; Flávio Teles, MD, PhD, Principal Investigator — Universidade Estadual de Ciências da Saúde de Alagoas; Rogério Passos, Principal Investigator — Hospital São Rafael S.A
Locations (1):
- Marcelo Augusto Duarte Silveira, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teles F, da Silva TM, da Cruz Junior FP, Honorato VH, de Oliveira Costa H, Barbosa AP, de Oliveira SG, Porfirio Z, Liborio AB, Borges RL, Fanelli C. Brazilian red propolis attenuates hypertension and renal damage in 5/6 renal ablation model. PLoS One. 2015 Jan 21;10(1):e0116535. doi: 10.1371/journal.pone.0116535. eCollection 2015. PMID 25607548
- [Background] Dai L, Golembiewska E, Lindholm B, Stenvinkel P. End-Stage Renal Disease, Inflammation and Cardiovascular Outcomes. Contrib Nephrol. 2017;191:32-43. doi: 10.1159/000479254. Epub 2017 Sep 14. PMID 28910789
- [Result] Silveira MAD, Teles F, Berretta AA, Sanches TR, Rodrigues CE, Seguro AC, Andrade L. Effects of Brazilian green propolis on proteinuria and renal function in patients with chronic kidney disease: a randomized, double-blind, placebo-controlled trial. BMC Nephrol. 2019 Apr 25;20(1):140. doi: 10.1186/s12882-019-1337-7. PMID 31023272
- [Result] Cobo G, Lindholm B, Stenvinkel P. Chronic inflammation in end-stage renal disease and dialysis. Nephrol Dial Transplant. 2018 Oct 1;33(suppl_3):iii35-iii40. doi: 10.1093/ndt/gfy175. PMID 30281126
- [Derived] Duarte Silveira MA, Malta-Santos H, Reboucas-Silva J, Teles F, Batista Dos Santos Galvao E, Pinto de Souza S, Dantas Dutra FR, Dantas Gomes MM, Teixeira MB, Miranda Rebelo da Conceicao LF, Nascimento CS, Vasques Nonaka CK, Cezar RS, Pena Batista PB, Berretta AA, Borges VM, da Hora Passos R. Effects of Standardized Brazilian Green Propolis Extract (EPP-AF(R)) on Inflammation in Haemodialysis Patients: A Clinical Trial. Int J Nephrol. 2022 Nov 22;2022:1035475. doi: 10.1155/2022/1035475. eCollection 2022. PMID 36457860